CLINICAL TRIAL: NCT02482363
Title: UVA Irradiation of Skin in Pregnant Women Increases Uterine Artery Blood Flow and Reduces Blood Flow Through a Nitric Oxide Pathway
Brief Title: Vascular Responses to UV Exposure in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 170108
Record Dates: First submitted 2015-06-12; First posted 2015-06-26 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active UVA radiation (Active Comparator): This arm will receive 20 minutes of UVA to the skin while resting quietly.
  Interventions: Radiation: UVA radiation
- Sham control (Sham Comparator): This arm will receive 20 minutes of quiet rest and heat but with their skin protected from UVA
  Interventions: Radiation: Sham Control

INTERVENTIONS:
Radiation: UVA radiation — 20 minutes of low dose UVA from a phototherapy unit
  Arms: Active UVA radiation
Radiation: Sham Control — 20 minutes of sham control exposure
  Arms: Sham control

SUMMARY:
Season of birth influences pregnancy for reasons that remain unclear however the answer may lie in the amount of sunshine pregnant women are exposed to. Sunshine, or ultraviolet light (UV) exposure is already known to have benefits for health on heart disease, strokes and depression. In pregnancy, relationships between sunshine exposure are evident in birth weight, preterm birth and risk of blood pressure complications. Vitamin D, the UV generated hormone, was thought to be responsible when low vitamin D levels were associated with these pregnancy complications. However, vitamin D replacement is ineffective at preventing these outcomes, and the investigators hypothesise that this is because it is the UV that is beneficial for pregnancy and it is working through a different pathway.

A new understanding of skin function is central to this, with a 2014 study showing that exposing an adult to 20 minutes of low dose UV light lowered their blood pressure and improved blood flow. These investigators demonstrated this was a direct effect of UV on the skin and was mediated by nitric oxide, a chemical central to many aspects of pregnancy including blood pressure regulation and uterine activity.

The investigators in this study have funding from Tommy's to investigate if a similar effect is seen in pregnancy on the circulation. The design is similar to the previously successful method and volunteers would be recruited from clinical areas during the second trimester. As both resting and warming for 20 minutes have the potential to have similar effects on the circulation, a control arm will expose participants to these without the UV.

This pilot study would involve one visit and measurements taken would include heart rate, blood pressure, arteriography, ultrasound of the uterine arteries and blood measurements of nitric oxide levels. Arteriography is performed using a specialised arm cuff and is safe and non-invasive. A subset of these women would be invited to repeat this in the third trimester to investigate for a difference in effect at a later gestation.

DETAILED DESCRIPTION:
The hypothesis is that ultraviolet A (UVA) exposure during pregnancy will release nitric oxide (NO) from the skin and that in turn this will cause blood vessel dilatation. This will be seen by changes in uterine artery blood flow, blood pressure, and arterial stiffness (arteriography). The aim is to investigate this in a low risk group and a high risk group, as these 2 groups of women have different baseline characteristics of their vascular system and potentially different responses to our intervention. A subset of these women will be invited to repeat the intervention in the third trimesters of their pregnancies to establish if the effect differs with advancing gestation. Birth outcomes on participants will be collected to check if the high and low risk groups are representative of this status.

Participant contact information will be kept separately from their collected data to anonymise the collected data and all outcome data will be de-identified. All collected information will be stored on secure university servers that are password protected.

Participants will be recruited to participate in the low sunshine months November 1st until March 1st to minimise background sunshine and UV exposure.

LOW RISK ARM:

20 participants will be recruited from community and hospital antenatal clinics, day assessment unit, labour ward or at first trimester screen appointment by posters, a research midwife or a member of clinical research team. Potential participants will be given an information form and will be asked to give written consent following sufficient time for consideration.

The participants will be between 14 and 28 weeks pregnant at the time of the intervention and have no pregnancy related complications or risk factors for pre-eclampsia or growth restriction.

Over a single morning or afternoon the protocol will be completed with the participant exposed to both the intervention and the control in the one 4 hour period. The intervention participants will be exposed to is ultraviolet A for 20minutes in a dermatology phototherapy cabinet. This is the equivalent of 2 standard erythemal doses (SED's) of UV light exposure. On a normal summer day in Northern Europe the general population would expect to receive 30-40 SED's. In the control intervention participants will be exposed to sham irradiation where they will undergo this exposure while wearing a loose fitting paper boiler suit that is UVA impenetrable to prevent UVA exposure. Protective sunglasses will be provided.

On arrival at the Wellcome Trust Clinical Research Facility, participants will be randomized to the active or control treatment arm first with a simple randomisation method (coin toss) by a member of the clinical research team. As the groups will be controlled for risk factors, the main important covariate is age. The purpose of randomisation in this setting is to aid with blinding the ultrasound investigator to which arm the patient is in, as the investigator can affect ultrasound results. As such, a simple randomisation procedure such as a coin toss by the research nurse on arrival is appropriate. One toss will determine group allocation with heads getting control exposure first and tails getting intervention first. This will be recorded on the participant information sheet and unblinded for analysis. The participant will then rest seated for 30 minutes in comfortable clothing in a temperature controlled room at 25 degrees Celsius. They will be assigned a study number and the researcher will collect pregnancy and maternal characteristics.

A member of the research team will measure baseline blood pressure, skin temperature, heart rate and perform arteriography. Arteriography has a standard collecting procedure and is an established tool to measure stiffness of the aorta (the largest blood vessel from the heart). An ultrasound will confirm fetal viability and baseline uterine artery Doppler measurements. An intravenous (IV) cannula will be inserted and a 5ml venous blood sample will be collected by an experienced member of the clinical research team.

The participant will then be exposed to the intervention of UVA for 20 minutes in either their underwear (active) or in a loose fitting paper boiler suit that is UVA impenetrable. The suit allows the skin to heat up, but not be exposed to the UVA. This controls for any temperature effects. The investigator performing ultrasound is blinded to whether the participant was wearing the suit or not by the use of a research nurse and the investigator not being present during the irradiation.

Immediately following exposure BP, heart rate, skin temperature and uterine artery Doppler's will be measured at 10 minutely intervals for 1 hour. 3 measurements will be collected at each time point for BP, heart rate and uterine artery Doppler. A venous blood sample will be collected from the cannula at the 0, 30 and 60 minute time points. At the 60 minute time point, arteriography will be repeated. Uterine artery Doppler images will be stored with a study number for offline analysis.

The participant will then cross over in to the other arm, which the investigator remains blind to and the process is repeated.

HIGH RISK ARM:

20 participants between 14 and 28 weeks will be referred from their direct care team based on historical risk factors in a previous pregnancy or high risk factors in their current pregnancy including essential hypertension, renal or vascular disease, previous intrauterine growth restriction or from a low Papp-A result on their first trimester screening blood tests. Papp-A is measured as part of first trimester screening and is produced by the developing placenta. Low results are associated with poor fetal growth and pre-eclampsia. Their direct care team in community or hospital antenatal clinics, day assessment unit or in the ultrasound department may identify these potential participants and refer them to the research team if they are interested in participating. This will include midwives, doctors and ultrasound staff. A poster and mechanism for self referral will be present in the care areas of antenatal clinic and the ultrasound department. If they give consent, they will be recruited to participate. If there is any concerns about fetal or maternal well being they will be excluded from this trial.

They will undergo the above protocol including randomisation.

LONGITUDINAL ARM:

All participants will be invited to return to undergo the trial protocol again at a third trimester time point within the 3 month window that the trial is being run. The investigators would aim to collect 10 from the low risk group and 10 from the high risk group. Participants whose third trimester commences outside this window will not be eligible for the longitudinal group.

FOR ALL GROUPS:

The consent will include permission to collect birth outcomes once they are delivered. Outcomes of interest will be pregnancy outcome (stillbirth, live birth), birth weight, gestational length, incidence of pre-eclampsia or pregnancy induced hypertension. This will be retrieved from the medical record and will be used for post hoc subgroup analysis to assess for any difference in response to UVA exposure. The study will conclude once the last baby is delivered and their birth data collected.

Results will be recorded in an anonymised way with a study number, and anonymised data will be stored separately to participant data. After the last pregnancy is delivered, all data will be completely de-identified. Blood samples will be stored in the Edinburgh Reproductive Tissue Biobank with participant consent.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant volunteers
* Ages 18- - 45
* No significant medical or obstetric history
* English speaking
* Able to provide informed consent
* Singleton pregnancy
* Low risk first trimester screen
* Have 4 hours of time
* Historical risk factors for growth restriction or pre-eclampsia
* Papp A < 0.40 MoMs

Exclusion criteria:

* Non english speaking
* Smoking
* History of intrauterine growth restriction (IUGR) or pre-eclampsia
* BMI >40
* Contraindication to UV exposure
* History of blood born viruses (hepatitis B, C, HIV)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Uterine artery Doppler | Change over 60 minutes following exposure
  The uterine artery will be interrogated with abdominal ultrasound to determine diameter and Doppler measurements to calculate resistance indices (PI) and flow velocity. This will be done at baseline and at 10 minutely intervals following exposure for 60 minutes.

SECONDARY OUTCOMES:
Blood pressure | 60 minutes
  Blood pressure will be measured with an appropriate sized cuff to determine blood pressure at baseline and the at ten minutely intervals following exposure.
Nitrospecies | 60 minutes
  Nitrate and nitrite levels will be measured in the venous circulation at baseline. These are metabolites of nitric oxide metabolism.
Arteriography | 60 minutes
  Arteriography is a measurement that reflects changes in air

CONTACTS AND LOCATIONS:
Overall Officials: SARAH STOCK, BSc MBChB, Principal Investigator — QUEEN'S MEDICAL RESEARCH INSTITUTE
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom